CLINICAL TRIAL: NCT05719376
Title: The Effect of Intravenous Iron Therapy and Erythropoiesis-stimulation Agent Combination on Renal Transplant Outcomes
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-1314
Record Dates: First submitted 2023-01-18; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: Monofer (experimental)
- control (Other): Follow the criteria for investigational product
  Interventions: Drug: control group

INTERVENTIONS:
Drug: Monofer (experimental) — Monofer 200mg : OP-28day, OP-21day, OP-7day, OP day, POD #7 IV injection, Mircera 120mcg SQ : OP-7 day~OP-1day
  Arms: Experimental
Drug: control group — Ferritin<100, TSAT<20 : Monofer 200mg IV, twice/ Ferritin 100~200, TSAT<20 : Monofer 200mg IV, once / Ferritin 201~500, TSAT<20 : Monofer 100mg IV, once / Not administer in any other case
  Arms: control

SUMMARY:
RBC transfusion (RBCT) after kidney transplantation(KT) is about 50%. Anemia is common after kidney transplant surgery due to intraoperative blood loss, delayed graft function, and side effects of immunosuppressive drugs. However, due to exposure to non-self human leukocyte antigens (HLA) from blood transfusion, there is a risk of sensitization to HLA through the production of anti-HLA antibodies. In renal transplant patients, exposure to non-self HLA antigens due to RBCT can lead to the generation of donor-specific antibodies (DSA) against renal allograft donors. Patients who have undergone KT are frequently exposed to RBCT, and immunologic damage resulting from this can be an important cause of loss of graft kidney function. Therefore, there should be a more careful review of the risk associated with RBCT on KT recipients.

Of the 16,191 Koreans who underwent KT between 2008 and 2017, 59.7% received transplant-related blood transfusions. As a result of analyzing 13,871 Koreans who underwent KT between 2007 and 2015, the overall graft failure rate was 15.5%, and the hazard ratio of survival rate according to RBCT before and after KT increased as the amount of transfusion increased. RBCT before and after KT was independently associated with graft failure and death. Therefore, research on treatment methods that can effectively reduce blood transfusion in transplant patients is absolutely necessary. About 30-60% of patients undergoing major surgery show preoperative anemia, which causes blood transfusions, complications during hospitalization, prolonged hospitalization, and delayed recovery. The most common cause of anemia is iron deficiency. In particular, an increase in hepcidin, a major regulator of iron metabolism, reduces intestinal iron absorption and promotes iron sequestering by macrophages, resulting in a state of functional iron deficiency. Therefore, oral iron intake as a treatment for anemia in surgical patients is not effective. Although the safety and clinical superiority of high-dose intravenous iron therapy have been demonstrated in patients with chronic renal failure, the effect of this drug on blood transfusion of pre- and post-kidney transplant surgery has not been studied. Therefore, this study aims to verify the effectiveness and stability of the combined administration of intravenous(IV) iron and erythropoiesis-stimulating agents(ESA) before and after KT for patients who perform KT for end-stage kidney disease(ESKD). The investigators will analyze hemoglobin, transferrin saturation, ferritin changes, and transfusion requirements according to the combined administration of IV iron and ESA before and after surgery of kidney transplant patients. Also, the investigators evaluate whether a treatment combining IV iron and ESA will be possible as an alternative blood transfusion treatment and its effect on the clinical prognosis of KT recipients. In particular, the effect on the function of the graft kidney, immunological outcomes-DSA, antibody-mediated rejection, and survival rate will be analyzed. Also, the investigators will analyze the change in expression of hepcidin and oxidative stress markers before and after kidney transplantation and the mechanism of expression according to the combined administration of IV iron and ESA. This study is a multicenter(including 3 centers), open-label, prospective, and randomized clinical trial. 302 patients undergoing living-donor KT for ESKD are randomly assigned in a 1:1 ratio to an experimental group actively using IV iron and ESA, and a control group receiving conventional anemia treatment for 42 months from the time of IRB approval. Participants selected for the experimental group will be given a total of 1000 mg of IV Monofer(iron isomaltoside); each 200 mg dose on 28, 21, and 7 days before kidney transplantation, on the day of surgery, and 7 days after surgery. In the case of ESA, it is freely used according to the criteria up to 7 days before transplantation and subcutaneously injected with 120 mcg of Mircera(methoxy polyethylene glycol-epoetin beta) between 7 days before surgery and a day before surgery. In the control group, IV Monofer is administered only 28 days before surgery according to the set criteria. Mircera is also freely used in the control group according to the criteria up to 7 days before KT but not used between 7 days before surgery and a day before surgery.

DETAILED DESCRIPTION:
Total 302 subjects, Experimental group vs Control group, 1. Experimental group :

* Total of 1000 mg Monofer(iron isomaltoside) IV injection; each Monofer 200mg dose on ①28, ②21, and ③7 days before KT,

  * on the day of surgery, and ⑤7 days after surgery
* Mircera(methoxy polyethylene glycol-epoetin beta) 120mcg SQ once : between 7 days before surgery and a day before surgery.

  * In the case of ESA, it is freely used according to the criteria up to 7 days before transplantation

  2. Control group :at 28 days before KT, Monofer is administered according the following criteria.
* Ferritin <100 μg/L & TSAT<20% : Monofer 200mg IV, twice
* Ferritin 100~200 μg/L & TSAT<20% : Monofer 200mg IV, once
* Ferritin 201~500 μg/L & TSAT<20% : Monofer 100mg IV, once
* Not administer in other cases * In the case of ESA, it is freely used according to the criteria up to 7 days before transplantation

ELIGIBILITY:
Inclusion Criteria:

1. living donor transplantation (age>19)
2. Ferritin<700㎍/L, TSAT<40%

Exclusion Criteria:

1. CDC(+), FXM(+)
2. Active infection
3. Hematologic malignancy, monoclonal gammaglobulin Dz, Hematologic Dz induced anemia
4. Receiving treatment of malignant tumor
5. HIV (+)
6. ALT, AST > 3 times upper limit of normal

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the number of blood transfusions according to the combination of intravenous iron therapy and EPO agent on perioperative period | From 1 month before operation to 1 year after operation (28 days before operation, 1st day, 10th day, 1month, 12month after operation)
  Comparison of the number of blood transfusions(packed RBC transfusion) according to the combination of intravenous iron therapy and EPO agent on perioperative period

SECONDARY OUTCOMES:
comparison of changes in anemia parameters(ferritin in ng/mL) | From 1 month before operation to 1 year after operation(28 days before operation, 1st day, 10th day, 1month, 12month after operation)
  comparison of changes in anemia parameters(ferritin in ng/mL)
comparison of changes in anemia parameters(TSAT in %) | From 1 month before operation to 1 year after operation(28 days before operation, 1st day, 10th day, 1month, 12month after operation)
  comparison of changes in anemia parameters(TSAT in %)
comparison of changes in anemia parameters(EPO level in mU/mL) | From 1 month before operation to 1 year after operation(28 days before operation, 1st day, 10th day, 1month, 12month after operation)
  comparison of changes in anemia parameters(EPO level in mU/mL)
comparison of changes in hepcidin expression level in pg/mL | From 1 month before operation to 1 year after operation(28 days before operation, 1st day, 10th day, 1month, 12month after operation)
  comparison of changes in hepcidin expression level in pg/mL
comparison of changes in oxidative stress marker | From 1 month before operation to 1 year after operation(28 days before operation, 1st day, 10th day, 1month, 12month after operation)
  comparison of changes in oxidative stress marker(MDA in mmol/L, 4-HNE in pg/mL, NGAL in ng/mL)
comparison of changes in immunologic parameters following the administration of intravenous iron therapy and EPO agent | From 1 month before operation to 1 year after operation(28 days before operation, 1st day, 10th day, 1month, 12month after operation)
  comparison of changes in immunologic parameters(de novo DSA in MFI, antibody-mediated rejection rate in %, death censored graft survival and patient survival rate in %) following the administration of intravenous iron therapy and EPO agent

CONTACTS AND LOCATIONS:
Overall Officials: Kyu ha huh, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No